CLINICAL TRIAL: NCT03380351
Title: The Implementation of Cognitive Screening and Educational Support to Improve Outcomes of Adolescents and Young Adults With Sickle Cell Disease: From Clinic to the Community and Back
Brief Title: Specifying Interventions From the Sickle Cell Disease Implementation Consortium (SCDIC)
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 3U01HL133994-02S1 (NIH); 3U01HL133994-02S1 (NIH)
Record Dates: First submitted 2017-11-20; First posted 2017-12-21 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Anemia, Sickle Cell
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SCDIC interventions: Careful detail the intervention components and the implementation strategies (i.e., the mechanisms by which the interventions are being delivered in usual care) being developed by the consortium.
  Interventions: Behavioral: SCDIC interventions

INTERVENTIONS:
Behavioral: SCDIC interventions — The research team will characterize the intervention components and their implementation strategies.

SUMMARY:
The goal of this study is to specify the interventions, implementation strategies and control conditions from the Sickle Cell Disease Implementation Consortium (SCDIC) using a mixed-methods approach to study site materials and conduct semi-structured qualitative interviews with site representatives (N=3 per site). We focused on the Emergency Department Working Group from the SCDIC working groups.

DETAILED DESCRIPTION:
The long-term goal of this line of research is to identify the most effective components of SCD interventions while also identifying effective implementation strategies informed by a systematic and rigorous work done by the members of the SCDIC consortium to improve the quality of life of people with SCD, a life-threatening hematological disorder. This study aims to collect detailed information about the planned interventions, the implementation strategies and the control conditions from each site.

ELIGIBILITY:
Inclusion Criteria:

* three representatives of each of the SDIC sites: the Principal Investigator, and two people nominated by the PI.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is focused on gathering data about the interventions planned and delivered from three different stakeholders of each site.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
SCDIC Framework of Interventions | 2 years
  Detailed descriptions of the interventions being developed by the SCDIC including a) entity, or entities, targeted by the intervention; (b) functional domains targeted by the interventions; and (c) delivery system characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Ana Baumann, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Along the study, we will share the information gathered with participants to check for accuracy. The framework of the interventions will be shared with the participants during the SCDIC Steering Committee calls.
Supporting Information: Study Protocol, ICF
Time Frame: data will be available in two years for the remaining of the 2 years of the consortium.
Access Criteria: Assess will be given to all participants via the Consortium's webpage
URL: https://scdic.rti.org/

REFERENCES:
- [Derived] Nwosu C, Khan H, Masese R, Nocek JM, Gollan S, Varughese T, Bourne S, Clesca C, Jacobs SR, Baumann A, Klesges LM, Shah N, Hankins JS, Smeltzer MP. Recruitment Strategies in the Integration of Mobile Health Into Sickle Cell Disease Care to Increase Hydroxyurea Utilization Study (meSH): Multicenter Survey Study. JMIR Form Res. 2024 Apr 16;8:e48767. doi: 10.2196/48767. PMID 38625729
- [Derived] Baumann AA. Commentary: Adapting and Operationalizing the RE-AIM Framework for Implementation Science in Environmental Health: Clean Fuel Cooking Programs in Low Resource Countries. Front Public Health. 2020 Jun 9;8:218. doi: 10.3389/fpubh.2020.00218. eCollection 2020. No abstract available. PMID 32582613
- [Derived] Baumann AA, Belle SH, James A, King AA; Sickle Cell Disease Implementation Consortium. Specifying sickle cell disease interventions: a study protocol of the Sickle Cell Disease Implementation Consortium (SCDIC). BMC Health Serv Res. 2018 Jun 27;18(1):500. doi: 10.1186/s12913-018-3297-1. PMID 29945631